CLINICAL TRIAL: NCT00970554
Title: Effectiveness of Telescopic Magnification in the Treatment of Amblyopia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Agnes Wong, Ophthamologist-In-Chief, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000011712
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Amblyopia
Keywords: Amblyopia; Telescopic magnification; Patching
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patching only (Active Comparator)
  Interventions: Other: Patching
- Patching plus telescope group (Experimental)
  Interventions: Other: Telescopic magnification

INTERVENTIONS:
Other: Patching — Patching of the sound eye for 30 minutes a day for 17 weeks.
  Arms: Patching only
Other: Telescopic magnification — Patching of the sound eye plus simultaneous use of a telescopic device by the amblyopic eye for 30 minutes a day for 17 weeks.
  Arms: Patching plus telescope group

SUMMARY:
Amblyopia is a visual impairment of one eye that results from disuse of that eye during early brain development. The standard treatment for amblyopia consists of patching or pharmacological penalization of the sound eye. Unfortunately, approximately 50% of amblyopic children do not respond to these therapies, with poor compliance being a major factor in treatment failure. One new treatment strategy involves patching the sound eye while using a telescopic device on the amblyopic eye to magnify the images formed in the amblyopic eye. Children were randomized to receive either daily patching of the sound eye for 30 minutes only (patching only group), or daily patching of the sound eye for 30 minutes plus simultaneous use of a telescopic device by the amblyopic eye during patching (patching plus telescope group).

DETAILED DESCRIPTION:
The goal of the present investigation was to conduct a prospective randomized clinical study to further evaluate the effectiveness of telescopic magnification plus patching vs patching alone on different types of amblyopia in patients who had failed previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4-17 years
* Strabismic, refractive (anisometropic), isometropic or mixed mechanism amblyopia

  * Strabismic amblyopia is defined as amblyopia (1) in the presence of either an inability to maintain parallel visual axes (heterotropia) at distance or near fixation or both, or a history of strabismus surgery (or botulinum injection), and (2) in the absence of refractive error meeting the criteria below for mixed mechanism amblyopia
  * Refractive/Anisometropic amblyopia is defined as amblyopia in the presence of a difference in refractive error between the two eyes (anisometropia) of ≥0.5 diopter (D) of spherical equivalent or ≥1.5D of difference in astigmatism in any meridian, with no measurable heterophoria at distance or near fixation, which persisted after 12 weeks of spectacle correction
  * Isometropic amblyopia is defined as amblyopia in the presence a refractive error ≥5.0D of spherical equivalent in both eyes, but not meeting the criteria of anisometropic amblyopia
  * Mixed mechanism strabismic and refractive amblyopia is defined as the presence of both strabismic and anisometropic types of amblyopia
* Ability to read the ETDRS letter chart
* Visual acuity between 0.3 and 1.3 logMAR (i.e., between 20/40 and 20/400) in the amblyopic eye
* Visual acuity of 0.3 logMAR (i.e., 20/40) or better in the sound eye
* Interocular acuity difference ≥0.3 logMAR
* Appropriate refractive error correction for at least 12 weeks

Exclusion Criteria:

* Presence of an ocular cause of reduced visual acuity
* Myopia with a spherical equivalent of -6.0D or more, due to the likely presence of pathological myopia
* Prior intraocular surgery
* Known skin reaction to patch or bandage adhesive

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2007-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The best corrected logMAR visual acuity score of the amblyopic eye. | 17 weeks

SECONDARY OUTCOMES:
Visual acuity of at least 0.2 logMAR (20/30) and/or improvement of at least 0.2 logMAR from baseline in the amblyopic eye. | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Wong, MD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wu J, Nazemi F, Schofield J, Mirabella G, Wong AM. Effectiveness of telescopic magnification in the treatment of amblyopia: a pilot study. Arch Ophthalmol. 2010 Mar;128(3):297-302. doi: 10.1001/archophthalmol.2009.400. PMID 20212198